CLINICAL TRIAL: NCT02881281
Title: Development of Problem-solving Skills Among Female Adolescents by Application of Social Cognitive Theory in Parent-Child Relationship
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Payam Peymani, Director of Health Policy Research Center of Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SUMSUNIVERSITY
Record Dates: First submitted 2016-06-22; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Adolescent Girls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Other): Education program
  Interventions: Other: educational program for Development of problem-solving skills
- Control Group (Other): no intervention
  Interventions: Other: no education program

INTERVENTIONS:
Other: educational program for Development of problem-solving skills
  Arms: Education
Other: no education program — no education program
  Arms: Control Group

SUMMARY:
Adolescence is the most important period of growth for humans. The conflict and disagreement which exists within family relationships will affect the children behaviors. Family relationships are the cause of many problems in adolescents, to develop a training program on problem-solving skills for adolescent girls to change their relationship with their parents.

ELIGIBILITY:
Inclusion Criteria:

* female secondary schools
* healthy body,
* not having a psychiatric disorder

Exclusion Criteria:

* psychiatric disorder
* not being volunteer to participate in the present study.

Ages: 12 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Child-Parent Relationship. | 4 month
  In this study, will be reported changes in parent-child relationship with pre and post-test. This change will be measured by Child-Parent Relationship Scale (Fine et al, 1983) with the aim of evaluating the relationships between parent and child. This scale is a 24 question tool which has 4 sub-scales of positive affection, role confusion, replication, and relationship. This scale included a 7-item Likert. After the Farsi translation of this questionnaire, validity and reliability was confirmed among Iranian population by Sanaei (2009).
Constructs of social cognitive theory | 4 month
  In this study, will be reported changes in constructs of social cognitive theory (SCT) was developed by Bandura. Constructs of this hypothesis comprise knowledge and understanding of the position, expectations, values, self-efficacy, and self-regulation. This change will be measured by a researcher-made questionnaire based on the constructs of social cognitive theory to identify the knowledge and understanding of the position, expectancies, values, self-efficacy and self-regulation. In order to prepare this section of instruments, after a literature review on information resources, a questionnaire was designed. For determining the content validity of the tools, the questionnaires will be given to ten faculty members in the related subjects. In this study, will be reported changes in constructs of social cognitive theory (SCT) was developed by Bandura.

CONTACTS AND LOCATIONS:
Locations (1):
- Seyed Taghi Heydari, Shiraz, Fars, Iran